CLINICAL TRIAL: NCT01529632
Title: A Study to Compare the Efficacy and Safety of Once Daily QVA149 Versus the Once Daily Concurrent Administration of QAB149 Plus NVA237 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Comparison of Safety and Efficacy of the Combination Product QVA149A Against the Concurrent Administration of the Individual Components, QAB149 and NVA237, in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: BEACON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2326; 2011-006050-91 (EudraCT Number)
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; QVA149; QAB149; NVA237; indacaterol; glycopyrronium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Glycopyrrolate; indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 (Experimental): QVA149 plus placebo once daily for 28 days.
  Interventions: Drug: QVA149; Drug: Placebo
- QAB149 + NVA237 (Active Comparator): Indacaterol maleate (QAB149) plus glycopyrronium bromide (NVA237) once daily for 28 days.
  Interventions: Drug: NVA237; Drug: QAB149

INTERVENTIONS:
Drug: QVA149 — QVA149 110/50 ug supplied as capsules in blister packs for inhalation via SDDPI, once daily
  Arms: QVA149
Drug: NVA237 — NVA237 50 ug supplied as capsules in blister packs for inhalation via SDDPI, once daily
  Arms: QAB149 + NVA237
Drug: QAB149 — QAB149 150 ug supplied as capsules in blister packs for inhalation via SDDPI , once daily
  Arms: QAB149 + NVA237
Drug: Placebo — Placebo capsules provided in blister packs for inhalation via SDDPI, once daily
  Arms: QVA149

SUMMARY:
The study assessed the safety and efficacy of the fixed combination product QVA149 versus the component products QAB149 and NVA237, administered concurrently, in patients that have moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The study assessed the safety and efficacy of the fixed combination product QVA149 versus the component products QAB149 and NVA237, administered concurrently, in patients that have moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 40 yrs
* Smoking history of at least 10 pack years
* Diagnosis of COPD (moderate to severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2010)
* Post-bronchodilator FEV1 < 80% and ≥ 30% of the predicted normal value and post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion Criteria:

* Patients who have had a respiratory tract infection within 4 weeks prior to Visit 1
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular co-morbid conditions
* Patients with a known history and diagnosis of alpha-1 antitrypsin deficiency
* Patients in the active phase of a supervised pulmonary rehabilitation program
* Patients contraindicated for inhaled anticholinergic agents and β2 agonists

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Austria (4):
  - Novartis Investigative Site, Feldbach, Austria
  - Novartis Investigative Site, Grieskirchen, Austria
  - Novartis Investigative Site, Linz, Austria
  - Novartis Investigative Site, Wels, Austria
- Denmark (5):
  - Novartis Investigative Site, Aalborg, Denmark
  - Novartis Investigative Site, Hvidovre, Denmark
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Odense C
- Netherlands (8):
  - Novartis Investigative Site, Almelo, Netherlands
  - Novartis Investigative Site, Harderwijk, Netherlands
  - Novartis Investigative Site, Heerlen, Netherlands
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Hengelo
  - Novartis Investigative Site, Sittard-Geleen
  - Novartis Investigative Site, Tubbergen
  - Novartis Investigative Site, Veldhoven
- Norway (5):
  - Novartis Investigative Site, Kløfta
  - Novartis Investigative Site, Kongsvinger
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Trondheim
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uddevalla

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 193 patients were randomized, with 187 of those completing the study. A total of 6 patients discontinued from the study.
Pre-assignment Details: Open-label, active QAB149 and NVA237 were administered during a 14-day period prior to randomization in order to stabilize patients and standardize baseline lung function. The patients were then randomized to either the fixed dose combination or free combination arms of blinded treatment in a 1:1 ratio and received study drug for 28 days.
Groups:
- QAB149 + NVA237: Indacaterol (QAB149) plus glycopyrronium bromide (NVA237) once daily for 28 days.
Period: Overall Study
Arm/Group | QVA149 | QAB149 + NVA237
Started | 90 | 103
Completed | 87 | 100
Not Completed | 3 | 3
Not completed — Administrative problem | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | QAB149 + NVA237 | Total
Number analyzed (Participants) | 90 | 103 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (7.28) | 64.2 (7.40) | 64.9 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 44 | 76
  Male | 58 | 59 | 117

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) After 28 Days of Blinded Treatment
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 is defined as the average of the 23 hour 15 minute and 23 hour 45 minute post-dose FEV1 readings measured at day 29, after 28 days of treatment. Mixed model: Trough FEV1 = treatment + baseline FEV1 + FEV1 reversibility components + baseline smoking status + baseline ICS use + country + center (country) + error. Center was included as a random effect nested within country.
Time Frame: Day 29
Population: The Per Protocol Set includes the Full analysis Set patients with available data and without any major protocol deviations or criteria causing exclusion.
  Patients were analyzed according to the treatment to which they were randomized.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 + NVA237
Number analyzed (Participants) | 81 | 96
Liters | 1.459 (0.0196) | 1.465 (0.0180)

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) 0-4 Hours at Day 1
Description: Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) 0-4h at Day 1 was measured via spirometry conducted according to internationally accepted standards. Measurements were made at 0, 5, 15, and 30 minutes; and 1, 2, 3 and 4 hours post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. Mixed model used: AUC FEV1 = treatment + baseline FEV1 + FEV1 reversibility components + baseline smoking status + baseline ICS use + country + center (country) + error. Center was included as a random effect nested within country.
Time Frame: 0, 5, 15, and 30 minutes; and 1, 2, 3 and 4 hours post-dose at Day 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 + NVA237
Number analyzed (Participants) | 83 | 97
Liters | 1.597 (0.0125) | 1.573 (0.0114)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) 0-4 Hours at Day 28
Description: Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) 0-4h at Day 28 was measured via spirometry conducted according to internationally accepted standards. Measurements were made at 0, 5, 15, and 30 minutes; and 1, 2, 3 and 4 hours post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time. Mixed model used: AUC FEV1 = treatment + baseline FEV1 + FEV1 reversibility components + baseline smoking status + baseline ICS use + country + center (country) + error. Center was included as a random effect nested within country.
Time Frame: 0, 5, 15, and 30 minutes; and 1, 2, 3 and 4 hours post-dose at Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 + NVA237
Number analyzed (Participants) | 80 | 92
Liters | 1.575 (0.0200) | 1.587 (0.0184)

4. Secondary Outcome: Peak Forced Expiratory Volume in 1 Second (FEV1) on Days 1 and 28 Post-dose
Description: Spirometry was conducted according to internationally accepted standards. Peak FEV1 is the maximum FEV1 recorded in the period between 5 minutes and 4 hours post dose. Analysis of Covariance was carried out with a mixed model that used (period) baseline, defined as the value of FEV1 measured prior to the first study drug intake in the period, as a covariate.
Time Frame: 5 min - 4 hr at Days 1 and 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 + NVA237
Number analyzed (Participants) | 83 | 97
Liters
  Day 1 (n=83, 97) | 1.668 (0.0132) | 1.646 (0.0120)
  Day 28 (n= 80, 92) | 1.643 (0.0210) | 1.654 (0.0194)

5. Secondary Outcome: Time Course of Forced Expiratory Volume in One Second (FEV1) (Pre-dose to 4 Hours Post Dose) on Day 28
Description: Time course of Forced Expiratory Volume in 1 second (FEV1) was measured at -45 min, -15 min predose, 5 min, 30 min, 1 hr, 2hr, 3hr and 4 hr post-dose on Day 28. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: -45 min, -15 min predose, 5 min, 30 min, 1 hr, 2hr, 3hr and 4 hr post-dose on Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 + NVA237
Number analyzed (Participants) | 78 | 91
Liters
  -45 min predose (n=76,90) | 1.452 (0.0197) | 1.460 (0.0184)
  -15 predose (n=72,87) | 1.449 (0.0239) | 1.430 (0.0227)
  5 min postdose (n=76,89) | 1.491 (0.0222) | 1.514 (0.0206)
  30 min postdose (n=76,88) | 1.529 (0.0181) | 1.544 (0.0166)
  1 hour postdose (n=77,90) | 1.584 (0.0204) | 1.604 (0.0189)
  2 hours postdose (n=77,90) | 1.601 (0.0219) | 1.624 (0.0203)
  3 hours postdose (n=78,91) | 1.576 (0.0211) | 1.587 (0.0195)
  4 hours postdose (n=77,84) | 1.554 (0.0236) | 1.556 (0.0228)

6. Secondary Outcome: Change From Baseline in the Mean Daily, (Daytime and Nighttime Combined) Number of Puffs of Rescue Medication Used Over 28 Days of Treatment
Description: The number of puffs of rescue medication taken in the previous 12 hours was recorded in the Patient Diary in the morning and evening. The total number of puffs of rescue medication per day over the whole active treatment period was calculated and divided by the total number of days with non-missing rescue data to derive the mean daily number of puffs of rescue medication taken for the patient. If the number of puffs was missing for part of the day (either morning or evening) then a half day was used in the denominator.
Time Frame: Baseline and 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | QVA149 | QAB149 + NVA237
Number analyzed (Participants) | 84 | 95
puffs
  Baseline (day 1) | 2.24 (2.437) | 2.04 (2.585)
  28 days after treatment | 1.85 (2.283) | 1.70 (2.338)

7. Secondary Outcome: Change From Baseline in Percentage of Days With 'no Daytime Symptoms' Over 28 Days of Treatment
Description: The mean total symptom scores and mean individual symptom scores for the patient were calculated for the whole study period. The mean change from baseline in the total scores and in the individual scores were summarized by treatment and were analyzed for the percentage of 'nights with no nighttime awakenings'. The symptom variables for the whole active treatment period was analyzed using the similar MIXED model as for the primary endpoint, with the baseline FEV1 term being replaced by the respective baseline symptom variables.
Time Frame: 28 days
Population: The Modified per protocol set (PPS) was defined post-DBL and included all patients with available data and without any major protocol deviations or criteria or GCP finding causing exclusion. Patients were analyzed according to the treatment to which they were randomized.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | QVA149 | QAB149 + NVA237
Number analyzed (Participants) | 82 | 93
percentage of days
  Baseline (day 1) | 6.2 (16.54) | 3.9 (10.44)
  After 28 days of treatment | 9.3 (23.69) | 6.0 (15.85)

ADVERSE EVENTS:
Time Frame: From day 1 to day 28 and additional 30 days follow up.
Description: Safety Set included all patients who received at least one dose of study drug whether or not they were randomized.
Arm/Group | QVA149 | QAB149 + NVA237
Serious Adverse Events (participants affected / at risk) | 4/90 | 6/103
Other Adverse Events (participants affected / at risk) | 20/90 | 12/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=90) | QAB149 + NVA237 (N=103)
Pericarditis (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=90) | QAB149 + NVA237 (N=103)
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Oedema mouth (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 2 | 0
Influenza (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 7 | 6
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.